CLINICAL TRIAL: NCT04481126
Title: Acute Renal Insufficiency (ARI) Rate and Predictive Score of ARI in Hospitalized Patients for Acute Coronary Syndrome With ST-segment Elevation Needing Urgent Coronarography
Acronym: COROAKI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201021
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Acute Renal Insufficiency; Acute Coronary Syndrome
Keywords: Acute Renal Insufficiency; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Kidney Injury; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study aims to evaluate frequence of acute renal insufficiency in patients with ST-segment elevation who need urgent coronary angiography in Ambroise Paré hospital.

The secondary objectives are:

* identify factors of risks associated with the occurrence of acute renal insufficiency after coronarography.
* establish a preprocedure score, predicting of acute renal insufficiency after urgent coronary angiography in patients with ST+ acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patient aged ≥ 18 years;
* evocative symptoms of myocardiac ischemia: typical chest pain; ST-segment elevation and 1 mm in two consecutive peripheral leads and 2 mm in two consecutive precordial derivations, or appearance of a bloc of left branch of novo;
* need urgent coronarography;
* Covered by french social security scheme included CMU.

Exclusion Criteria:

* dialysed patient for chronic renal insufficiency;
* cardio-resporatory arrest;
* cardiogenic choc state;
* prior emergency passage to hospital;
* patient under tutor, gardianship;
* patient covered by french AME scheme;
* pregnant women or breastfeeding;
* all medical, psychological or social situation which should influents the compliance to protocol according to investigator;
* patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in Ambroise Paré hospital in the period between Jan 2017 to Jul 2019, who have been an urgent coronarography, and have a renal insufficiency needing dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
incidence of acute renal failure | at baselin and at 48 hours
  Acute renal failure is defined as an increase in plasma creatinine of at least 26.5µmol/l within 48 hours, or an increase in plasma creatinine of at least 1.5 times plasma creatinine within 48hours of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Paul GABARRE, MD, Principal Investigator — Nephrology department, Ambroise Paré hospital, APHP; Eve Vilaine, MD, Study Director — Nephrology department, Ambroise Paré hospital, APHP
Locations (1):
- Nephrology department, Ambroise Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No